CLINICAL TRIAL: NCT06566443
Title: Phase I Trial Evaluating the Safety of the Dietary Supplement Honokiol in Early-Stage Resectable Non-Small Cell Lung Cancer
Brief Title: Honokiol in Early-Stage Resectable Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Jun Zhang, Director of Thoracic Oncology, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PRO00037422 (HMCC-LU22-001)
Record Dates: First submitted 2024-08-09; First posted 2024-08-22 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — honokiol; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Honokiol (Experimental): Approximately, 15 patients will be enrolled in the study. They will take the study drug, honokiol, for 2 weeks prior to the surgery. The primary endpoint will be the maximum tolerated dose (MTD) of honokiol and this will be determined using Bayesian Optimal Interval Design (BOIN)
  Interventions: Drug: Honokiol

INTERVENTIONS:
Drug: Honokiol — Honokiol will be given orally at a starting dose of 1 capsule (250 mg/ capsule) per day for 2 weeks. Dose levels will escalate based on dose-limiting toxicity occurrence. We will start at one capsule (250 mg) once daily, dose 0 would be one capsule (250 mg) twice daily, dose +1 would be 500mg in the AM and 250mg in the evening, and +2 would be 500 mg twice daily.
  Other Names: Honopure (Dietary supplement)

SUMMARY:
This is a Phase I Trial evaluating the safety of the dietary supplement honokiol for lung cancer chemoprevention. Female or male patients aged 18 years, or older, with early stage lung cancer who have been scheduled for curative surgery will be eligible for participation in the study. The study will only enroll patients with stage I lung cancers less than 4 cm, given the recent approval of neoadjuvant chemotherapy and nivolumab for stage IB tumors > 4 cm. Approximately, 15 patients will be enrolled in the study. They will take the study drug, honokiol, for 2 weeks prior to the surgery. The primary endpoint will be the Maximum Tolerated Dose (MTD) of honokiol.

ELIGIBILITY:
Inclusion Criteria:

1. The patient provides written informed consent for the trial. Spanish speaking patients will be included and translation services will be provided as needed.
2. Male or female, 18 years of age or older, on the day of informed consent signing.
3. Early stage NSCLC eligible for upfront definitive surgical resection
4. Measurable disease according to the Response evaluation criteria in solid tumors (RECIST 1.1) within 30 days of treatment.
5. Expected life expectancy of at least 6 months
6. Adequate organ and marrow function as defined below:

   Hemoglobin ≥9.0 g/dl (without blood transfusion within 2 weeks of laboratory test used to determine eligibility) Absolute neutrophil count ≥1000/μL (without granulocyte colony stimulating factor support within 2 weeks of laboratory test used to determine eligibility) Platelet count ≥100,000/μL (without transfusion within 2 weeks of laboratory test used to determine eligibility)- Serum total bilirubin (TB) ≤1.5 x institutional upper limit of normal (ULN; In the case of known Gilbert's syndrome, a higher serum TB [>1.5 x ULN] is allowed), Aspartate transaminase/alanine transaminase ≤5 x institutional ULN Creatinine ≤1.5X the ULN or measured creatinine clearance ≥ 60 mL/min/1.
7. Willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits and examinations.

Exclusion Criteria:

1. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 3 weeks of trial treatment administration.
2. Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to trial treatment administration or who has not recovered (i.e., ≤ Grade 1 or at baseline) from Adverse Events (AEs) due to a previously administered agent.
3. Use of agents that target the mitochondrial metabolism.
4. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
5. The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
6. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
7. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
8. Eastern Cooperative Oncology Group (ECOG) performance status of ≥ 2.
9. Patients must have recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline. Patients with ≤ Grade 2 neuropathy may be eligible. If patient received major surgery, she must have recovered adequately from the toxicity and/or complications from the intervention prior to starting the trial treatment.
10. Active infection requiring systemic therapy.
11. Confirmed positive pregnancy test in women of childbearing potential (WOCBP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of Honokiol therapy | From treatment initiation of each patient, assessed up to 21 days after treatment initiation of final patient, up to 2 years after first enrollment.
  To determine the maximum tolerated dose (MTD) of honokiol therapy in patients with stage I NSCLC, less than 4 cm, who will undergo surgical resection. Review the safety data to determine the dose level at which the maximum tolerable level of toxicity is observed and select as the MTD the dose for which the isotonic estimate of the DLT rate is closest to the target DLT rate.

SECONDARY OUTCOMES:
Dose Limiting Toxicities of Honokiol therapy | DLT period will start with initial treatment dose until 21 days after.
  To determine the dose-limiting toxicity (DLT) and other toxicities associated with honokiol therapy, as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0;
Recommended Phase 2 Dose of Honokiol therapy | From initial treatment dose until 21 days after.
  To determine the recommended Phase II dose (RP2D) of honokiol; Bayesian Optimal Interval (BOIN) design will be used for dose finding.
Number of participants with tumor necrosis | From screening tissue collection to post-intervention tissue collection, an average of 3 months.
  To assess for any evidence of tumor necrosis.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | The safety period will start at baseline and will be assessed through study completion, up to 2 months
  To determine the safety and tolerability of honokiol therapy prior to surgery as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.

OTHER OUTCOMES:
Tissue immune correlative biomarkers of honokiol therapy | From pre-intervention blood collection to post-intervention blood collection, an average of 2 weeks.
  To evaluate tissue immune correlative biomarkers of honokiol therapy, including but not limited to Ki67, a good standard for the measurement of cell proliferation.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD, Principal Investigator — Houston Methodist Neal Cancer Center
Locations (1):
- Houston Methodist Neal Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Hsu PP, Sabatini DM. Cancer cell metabolism: Warburg and beyond. Cell. 2008 Sep 5;134(5):703-7. doi: 10.1016/j.cell.2008.08.021. PMID 18775299
- [Background] Barger JF, Plas DR. Balancing biosynthesis and bioenergetics: metabolic programs in oncogenesis. Endocr Relat Cancer. 2010 Sep 23;17(4):R287-304. doi: 10.1677/ERC-10-0106. Print 2010 Dec. PMID 20699334
- [Background] Cheng G, Zielonka J, Dranka BP, McAllister D, Mackinnon AC Jr, Joseph J, Kalyanaraman B. Mitochondria-targeted drugs synergize with 2-deoxyglucose to trigger breast cancer cell death. Cancer Res. 2012 May 15;72(10):2634-44. doi: 10.1158/0008-5472.CAN-11-3928. Epub 2012 Mar 19. PMID 22431711
- [Background] Liu H, Hu YP, Savaraj N, Priebe W, Lampidis TJ. Hypersensitization of tumor cells to glycolytic inhibitors. Biochemistry. 2001 May 8;40(18):5542-7. doi: 10.1021/bi002426w. PMID 11331019
- [Background] Kurtoglu M, Lampidis TJ. From delocalized lipophilic cations to hypoxia: blocking tumor cell mitochondrial function leads to therapeutic gain with glycolytic inhibitors. Mol Nutr Food Res. 2009 Jan;53(1):68-75. doi: 10.1002/mnfr.200700457. PMID 19072739
- [Background] Lampidis TJ, Bernal SD, Summerhayes IC, Chen LB. Selective toxicity of rhodamine 123 in carcinoma cells in vitro. Cancer Res. 1983 Feb;43(2):716-20. PMID 6848187
- [Background] Pathania D, Millard M, Neamati N. Opportunities in discovery and delivery of anticancer drugs targeting mitochondria and cancer cell metabolism. Adv Drug Deliv Rev. 2009 Nov 30;61(14):1250-75. doi: 10.1016/j.addr.2009.05.010. Epub 2009 Aug 27. PMID 19716393
- [Background] Chen F, Wang T, Wu YF, Gu Y, Xu XL, Zheng S, Hu X. Honokiol: a potent chemotherapy candidate for human colorectal carcinoma. World J Gastroenterol. 2004 Dec 1;10(23):3459-63. doi: 10.3748/wjg.v10.i23.3459. PMID 15526365
- [Background] Tsai TH, Chou CJ, Cheng FC, Chen CF. Pharmacokinetics of honokiol after intravenous administration in rats assessed using high-performance liquid chromatography. J Chromatogr B Biomed Appl. 1994 Apr 22;655(1):41-5. doi: 10.1016/0378-4347(94)00031-x. PMID 8061832
- [Background] Sporn MB, Suh N. Chemoprevention of cancer. Carcinogenesis. 2000 Mar;21(3):525-30. doi: 10.1093/carcin/21.3.525. PMID 10688873
- [Background] Lippman SM, Lee JJ, Sabichi AL. Cancer chemoprevention: progress and promise. J Natl Cancer Inst. 1998 Oct 21;90(20):1514-28. doi: 10.1093/jnci/90.20.1514. No abstract available. PMID 9790544
- [Background] Kelloff GJ, Sigman CC, Greenwald P. Cancer chemoprevention: progress and promise. Eur J Cancer. 1999 Dec;35(14):2031-8. doi: 10.1016/s0959-8049(99)00299-3. PMID 10711244
- [Background] Xu HL, Tang W, Du GH, Kokudo N. Targeting apoptosis pathways in cancer with magnolol and honokiol, bioactive constituents of the bark of Magnolia officinalis. Drug Discov Ther. 2011 Oct;5(5):202-10. doi: 10.5582/ddt.2011.v5.5.202. PMID 22466367
- [Background] Chiang CK, Sheu ML, Hung KY, Wu KD, Liu SH. Honokiol, a small molecular weight natural product, alleviates experimental mesangial proliferative glomerulonephritis. Kidney Int. 2006 Aug;70(4):682-9. doi: 10.1038/sj.ki.5001617. PMID 16807544
- [Background] Pan J, Zhang Q, Liu Q, Komas SM, Kalyanaraman B, Lubet RA, Wang Y, You M. Honokiol inhibits lung tumorigenesis through inhibition of mitochondrial function. Cancer Prev Res (Phila). 2014 Nov;7(11):1149-59. doi: 10.1158/1940-6207.CAPR-14-0091. Epub 2014 Sep 22. PMID 25245764
- [Background] Chen YJ, Wu CL, Liu JF, Fong YC, Hsu SF, Li TM, Su YC, Liu SH, Tang CH. Honokiol induces cell apoptosis in human chondrosarcoma cells through mitochondrial dysfunction and endoplasmic reticulum stress. Cancer Lett. 2010 May 1;291(1):20-30. doi: 10.1016/j.canlet.2009.08.032. Epub 2009 Oct 31. PMID 19880244
- [Background] Hahm ER, Singh SV. Honokiol causes G0-G1 phase cell cycle arrest in human prostate cancer cells in association with suppression of retinoblastoma protein level/phosphorylation and inhibition of E2F1 transcriptional activity. Mol Cancer Ther. 2007 Oct;6(10):2686-95. doi: 10.1158/1535-7163.MCT-07-0217. PMID 17938262
- [Background] Garcia A, Zheng Y, Zhao C, Toschi A, Fan J, Shraibman N, Brown HA, Bar-Sagi D, Foster DA, Arbiser JL. Honokiol suppresses survival signals mediated by Ras-dependent phospholipase D activity in human cancer cells. Clin Cancer Res. 2008 Jul 1;14(13):4267-74. doi: 10.1158/1078-0432.CCR-08-0102. PMID 18594009
- [Background] Crane C, Panner A, Pieper RO, Arbiser J, Parsa AT. Honokiol-mediated inhibition of PI3K/mTOR pathway: a potential strategy to overcome immunoresistance in glioma, breast, and prostate carcinoma without impacting T cell function. J Immunother. 2009 Jul-Aug;32(6):585-92. doi: 10.1097/CJI.0b013e3181a8efe6. PMID 19483651
- [Background] Tse AK, Wan CK, Shen XL, Yang M, Fong WF. Honokiol inhibits TNF-alpha-stimulated NF-kappaB activation and NF-kappaB-regulated gene expression through suppression of IKK activation. Biochem Pharmacol. 2005 Nov 15;70(10):1443-57. doi: 10.1016/j.bcp.2005.08.011. Epub 2005 Sep 21. PMID 16181613
- [Background] Deng J, Qian Y, Geng L, Chen J, Wang X, Xie H, Yan S, Jiang G, Zhou L, Zheng S. Involvement of p38 mitogen-activated protein kinase pathway in honokiol-induced apoptosis in a human hepatoma cell line (hepG2). Liver Int. 2008 Dec;28(10):1458-64. doi: 10.1111/j.1478-3231.2008.01767.x. Epub 2008 May 26. PMID 18507762
- [Background] Steinmann P, Walters DK, Arlt MJ, Banke IJ, Ziegler U, Langsam B, Arbiser J, Muff R, Born W, Fuchs B. Antimetastatic activity of honokiol in osteosarcoma. Cancer. 2012 Apr 15;118(8):2117-27. doi: 10.1002/cncr.26434. Epub 2011 Sep 20. PMID 21935912
- [Background] Hu H, Zhang XX, Wang YY, Chen SZ. Honokiol inhibits arterial thrombosis through endothelial cell protection and stimulation of prostacyclin. Acta Pharmacol Sin. 2005 Sep;26(9):1063-8. doi: 10.1111/j.1745-7254.2005.00164.x. PMID 16115372
- See also: Honokiol, magnolia bark, A miracle cure for cancer? — http://www.drchuang.com/honokiol-magnolia-bark-cancer-cure/
- See also: Bayesian Optimal Interval Designs for Phase I Clinical Trials — https://odin.mdacc.tmc.edu/~yyuan/Software/BOIN/paper.pdf